CLINICAL TRIAL: NCT04265924
Title: Increased FIO2 Influences SvO2 Interpretation and Accuracy of Fick-based Cardiac Output Assessment in Cardiac Surgery Patients
Brief Title: FIO2 Influences SvO2 Interpretation and Fick-based Cardiac Output Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-7177B
Record Dates: First submitted 2020-02-09; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Output

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- >0.85 FIO2 group (Active Comparator): This group receives FIO2 >0.85 during the surgery.
  Interventions: Other: fraction of inspired oxygen (FIO2)
- <0.7 FIO2 group (Active Comparator): This group receives FIO2 <0.7 during the surgery.
  Interventions: Other: fraction of inspired oxygen (FIO2)

INTERVENTIONS:
Other: fraction of inspired oxygen (FIO2) — The fraction of inspired oxygen (FIO2) is given accordingly (>0.85 for the >0.85 group, and <0.7 for the <0.7 group) to the patients during the surgery.

SUMMARY:
In this study, the investigators sought to clarify the influence of FIO2 levels on the variables in the Fick equation and then assessed the influence of each variable on the accuracy of Fick-CO measurements in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Patients who are aged ≥20 years, are undergoing planned elective cardiac surgery, and provided signed informed consent are included in the present study. Any patients with an intra-cardiac shunt are excluded.

The patients are randomly assigned to 2 groups: FIO2 <0.7 or FIO2 >0.85. And during the surgery, the oximeter values are kept ≥98%. Intra-operatively, FIO2, PaO2, SaO2, SvO2, PvO2, Hb, blood pH values, body temperature and TD-CO are recorded.

ELIGIBILITY:
Inclusion Criteria:

* undergoing planned elective cardiac surgery
* agree to sign informed consent

Exclusion Criteria:

* intra-cardiac shunt

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
The Hemoglobin Values in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will collect hemoglobin data in each patient.
The Oxygen Consumption in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will use the LaFarge equation to calculate oxygen consumption (ml/min/m^2) in each patient.
The Blood PH Values in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.
The Body Temperatures in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.
The SaO2 in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.
The SvO2 in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.
The PaO2 in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.
The PvO2 in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  The patients were divided into two FIO2 groups (FIO2 >0.85 or <0.7) during the surgery. We will calculate oxygen consumption in each patient.

SECONDARY OUTCOMES:
The Precision of Fick-based Cardiac Output in Different FIO2 Groups during Cardiac Surgeries | under general anesthesia but before surgical incision
  After collecting the elements data included in the Fick eqaution (oxygen consumption, hemoglobin, SaO2, SvO2, PaO2, and PvO2), we can calculate the Fick-based cardiac output in each patient. And the pulmonary artery thermodilution is adopted as the standard cardiac output monitoring method. We will calculate the correlation and level of agreement between Fick-based cardiac output and pulmonary artery thermodilution in the two groups.

REFERENCES:
- [Derived] Lin SY, Chang FC, Lin JR, Chou AH, Tsai YF, Liao CC, Tsai HI, Chen CY. Increased FIO2 influences SvO2 interpretation and accuracy of Fick-based cardiac output assessment in cardiac surgery patients: A prospective randomized study. Medicine (Baltimore). 2021 Sep 10;100(36):e27020. doi: 10.1097/MD.0000000000027020. PMID 34516492